CLINICAL TRIAL: NCT05433142
Title: A Phase 1 Multiple Dose Study to Evaluate the Safety and Tolerability of XmAb819 in Subjects With Relapsed or Refractory Clear Cell Renal Cell Carcinoma
Brief Title: Study of XmAb®819 in Subjects With Advanced Clear Cell Renal Cell Carcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Xencor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XmAb819-01
Record Dates: First submitted 2022-06-13; First posted 2022-06-27 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Clear Cell Renal Cell Carcinoma
Keywords: ccRCC; RCC; Renal Cell Cancer; Kidney Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation and Expansion (Experimental): Dose Escalation (Part A): Part A will establish the dosing schedule for XmAb819 administered IV and the dosing schedule of XmAb819 administered SC in subjects with ccRCC. The dosing schedule includes the priming dose, step-up priming dose(s), the minimum safe and biologically active dose.
  Dose Expansion (Part B): Part B-1 may administer XmAb819 IV, and Part B-2 may administer XmAb819 SC.
  Interventions: Biological: XmAb819

INTERVENTIONS:
Biological: XmAb819 — Monoclonal Bispecific Antibody

SUMMARY:
The purpose of this study is to assess the safety and tolerability of XmAb®819 administered intravenous (IV) or subcutaneous (SC) in subjects with relapsed or refractory clear cell renal cell carcinoma and to identify the minimum safe and biologically active dose and the recommended dose (RD).

DETAILED DESCRIPTION:
This is a Phase 1, multicenter, open-label, multiple-dose study designed in 2 parts: Part A, dose escalation, and Part B, dose expansion. The study is designed to establish the dosing schedule of XmAb819 administered IV and the dosing schedule of XmAb819 administered SC. The study is designed to evaluate safety and tolerability; to assess PK/PD and immunogenicity; and to preliminarily assess antitumor activity of XmAb819 in subjects with ccRCC. All eligible subjects will have relapsed or refractory disease after standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST 1.1) as assessed by the local site investigator. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Subjects who have relapsed and refractory ccRCC with evidence of disease progression on standard-of-care therapies
* ECOG performance status of 0 or 1.
* All subjects must have adequate tumor sample available (slides or archival FFPE blocks)

Exclusion Criteria:

* Prior treatment with an investigational anti-ENPP3/CD203c therapy
* History of serious allergic or anaphylactic/hypersensitivity reaction to monoclonal antibody therapy
* Systemic antineoplastic therapy within 5 half-lives on the first dose of study treatment.
* Failure to recover from any clinically significant toxicity related to previous anticancer treatment
* Have known active central nervous system metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are radiologically stable,
* Active known autoimmune disease (except that subjects are permitted to enroll if they have vitiligo; type 1 diabetes mellitus; residual hypothyroidism due to an autoimmune condition that is treatable with hormone replacement therapy only; psoriasis, atopic dermatitis, or another autoimmune skin condition that is managed without systemic therapy; or arthritis that is managed without systemic therapy beyond oral acetaminophen and nonsteroidal anti-inflammatory drugs)
* Evidence of any serious infection requiring IV anti-infective treatment within 14 days prior to the first dose of study drug
* Have a known additional malignancy that is progressing or has required active treatment within the past 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2022-06-13 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (safety and tolerability of XmAb819) | 28 days
  Safety and tolerability as assessed by incidence of TEAEs; incidence of clinically significant changes in safety laboratory tests, PE findings, vital signs, and ECGs; incidence and severity of CRS
Incidence of dose limiting toxicities (DLTs) | 28 days
  Safety and tolerability as assessed by incidence of DLTs and all available data which will be used to determine the optimal dose regimen.

SECONDARY OUTCOMES:
Measurement of Cmax | 56 days
  Peak plasma concentration (Cmax)
Measurement of AUCtau | 56 days
  Area under the plasma concentration versus time curve (AUCtau)
Objective Response rate | 42 days
  Objective response rate (RECIST 1.1 assessment of CT/MRI imaging)
Progression-free survival | 42 days
  Progression-free survival (RECIST 1.1 assessment of CT/MRI imaging)
Duration of response | 42 days
  Duration of response (RECIST 1.1 assessment of CT/MRI imaging)

CONTACTS AND LOCATIONS:
Overall Officials: Chet Bohac, MD, Study Director — Xencor, Inc.
Locations (8):
- United States (8):
  - Department of Medical Oncology and Therapeutics Research, City of Hope, Duarte, California
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - The University of Chicago Medical Center, Chicago, Illinois
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering, New York, New York
  - Duke University, Durham, North Carolina
  - Sarah Cannon Research Institute, LLC, Nashville, Tennessee
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No